CLINICAL TRIAL: NCT03973242
Title: Usefulness of Dual-focus Magnification With Narrow-band Imaging in the Prediction of Helicobacter Pylori Infection: a Prospective Randomized Trial
Brief Title: Dual-focus Magnification With Narrow-band Imaging in Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Wook Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DFHP2018
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Narrow Band Imaging

STUDY DESIGN:
Intervention Model Description: Study group: Dual Focus with Narrow band imaging Control group: White light endoscopy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DF-NBI (Active Comparator): Initially, gastric mucosa is observed by conventional wight light endoscopy. Then, converting to dual-focus mode with narrow band imaging is done. Gastric mucosa is observed once again by DF-NBI mode.
  Interventions: Device: Dual focus with narrow band imaging
- WL (Placebo Comparator): Conventional white light endoscopy use It is routine practice for the upper gastrointestinal endoscopy.
  Interventions: Device: Dual focus with narrow band imaging

INTERVENTIONS:
Device: Dual focus with narrow band imaging — dual focus mode for imaging magnification + narrow band imaging for the enhancement of mucosal vascularity and irregularity

SUMMARY:
Dual-focus with narrow-band imaging (DF-NBI) is a novel technique to improve the quality of images of the irregular mucosal structures and microvessels of gastric neoplasms. The investigators compare this technique with conventional white light (WL) endoscopy to predict Helicobacter pylori infection.

DETAILED DESCRIPTION:
The subjects are patients who underwent upper gastrointestinal endoscopy under sedation. Participants are randomized into DF-NBI and WL groups. Rapid urease test will be performed in all cases. By captured images of gastric mucosa, classification of DF-NBI for Helicobacter pylori infected mucosa will be developed and validated. The established classification of WL for Helicobacter pylori infection will be used. Finally, the investigators will compare the accuracy between two groups based on each classification.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients who have undergone uper gastrointestinal endoscopy for diagnosis or screening of cancer.

Exclusion Criteria:

* Those whose Hp status had already been clarified
* Pregnancy
* History of partial gastrectomy
* Taking proton pump inhibitor, antithrombotics or antibiotics within 4 weeks

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Accurate prediction of Helicobacter pylori status | 1 day
  Sensitivity, specificity, PPV, and NPV

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
If needed, IPD will be shared.